CLINICAL TRIAL: NCT05930665
Title: A Phase II, Prospective, Single Arm Trial of Cadonilimab in Combination With Bevacizumab and Standard Chemotherapy as First Line Therapy in Unresectable Pleural Mesothelioma
Brief Title: Study of Cadonilimab Combined With Bevacizumab and Standard Chemotherapy as First Line Therapy in Unresectable Pleural Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wenfeng Fang, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-028
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Pleural Mesothelioma
Keywords: bispecific antibody
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+Bevacizumab+Pemetrexed+Carboplatin (Experimental): Cadonilimab+Bevacizumab+Pemetrexed+Carboplatin for 4 to 6 cycles, followed by Maintenance with Cadonilimab and Bevacizumab
  Interventions: Drug: Cadonilimab+Bevacizumab+Pemetrexed+Carboplatin

INTERVENTIONS:
Drug: Cadonilimab+Bevacizumab+Pemetrexed+Carboplatin — Cadonilimab 10mg/kg intravenous (IV) every 3 weeks + Bevacizumab 7.5mg/kg IV every 3 weeks + Pemetrexed 500 mg/m² IV every 3 weeks + Carboplatin AUC 5 IV every 3 weeks for 4 to 6 cycles, followed by maintenance with Cadonilimab 10mg/kg IV every 3 weeks + Bevacizumab 7.5mg/kg IV every 3 weeks
  Other Names: AK104

SUMMARY:
Cadonilimab, a tetravalent bispecific antibody targeting PD-1 and CTLA-4, is designed to retain the efficacy benefit of combination of PD-1 and CTLA-4 and improve on the safety profile of the combination therapy. The aim of this study is to evaluate the efficacy and safety of cadonilimab in combination with bevacizumab and standard chemotherapy as first Line therapy in unresectable pleural mesothelioma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed pleural malignant mesothelioma not eligible for curative surgery
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
3. No previous systemic anti-tumor treatment for advanced/metastatic disease
4. Measurable disease as per mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.
5. Adequate haematological, renal and liver function.

Key Exclusion Criteria:

1. Primitive peritoneal, pericardial and tunica vaginalis testis mesothelioma.
2. Active, untreated central nervous system (CNS) metastasis.
3. Use of Chinese herbal medicine or immunomodulatory agents with anti-tumor indications within 14 days prior to the first dose of study treatment.
4. Known active autoimmune diseases.
5. Presence of other uncontrolled serious medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  defined as the percentage of participants who achieve a best overall response of complete response or partial response assessed according to mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 36 months
  defined as the time between the date of first dose of study drug and the date of first documented tumor progression per mRECIST v1.1, or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 36 months
  defined as the percentage of participants who achieve a best overall response of complete response, partial response, or stable disease assessed according to mRECIST v1.1 for assessment of response in malignant pleural mesothelioma.
Duration of Response (DoR) | Up to 36 months
  defined as the interval from the date of first documentation of objective response (complete response or partial response, according to the mRECIST v1.1) to the date of first documented tumor progression, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 36 months
  defined as the time between the date of first dose of study drug and the date of death due to any cause.
Adverse Events (AEs) | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China